CLINICAL TRIAL: NCT02361905
Title: Advantages of Ulipristal Acetate for the Preoperative Treatment of Hypoechoic Cellular Leiomyomas
Brief Title: Ulipristal Acetate for the Preoperative Management of Hypoechoic Cellular Leiomyomas
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Fulvio Zullo, Full professor, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UPA hypoecoic myomas
Record Dates: First submitted 2015-02-02; First posted 2015-02-12 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Fibroid
Keywords: fibroid; cellular leiomyomas; GnRH analogue; ulipristal acetate
MeSH Terms: conditions — Leiomyoma | interventions — ulipristal acetate; Leuprolide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ulipristal acetate (Experimental): women will be treated with an oral dose of ulipristal acetate 5 mg/day for 3 months
  Interventions: Drug: ulipristal acetate
- Leuprolile acetate (Active Comparator): Women will be treated with an intramuscular (IM) injection of leuprolide acetate 11.25 mg in the luteal phase
  Interventions: Drug: Leuprolide acetate

INTERVENTIONS:
Drug: ulipristal acetate — 5 mg/day will be administered starting from day 1 of the cycle and up to three months later
  Other Names: Esmya
  Arms: Ulipristal acetate
Drug: Leuprolide acetate — One dose of 11.25 GnRH analogue depot will be administered in the luteal phase of the menstrual cycle (days 21-24)
  Other Names: Enantone 11.25
  Arms: Leuprolile acetate

SUMMARY:
Cellular leiomyomas (CLs) are described as leiomyomas that are significantly more cellular than the surrounding myometrium, often with crowding and overlapping of nuclei. they often are soft and appear more tan or yellow and less circumscribed than the usual leiomyomas. Pre-operatively CLs can be recognized at ultrasound evaluation because they appear as hypoechoic uterine lesions. patients with hypoechoic myoma have a significantly longer surgery time after treatment with a gonadotropin-releasing hormone (GnRH) analog probably related to degenerative changes induced by this treatment. Hypoechoic CLs should be more responsive to ulipristal acetate treatment than common leiomyomas. The antiproliferative ulipristal effect, moreover, induces a condition of apoptotic necrosis that, compared to GnRH-a myxoid necrosis, probably allows an easier surgical enucleation of the tumor.

DETAILED DESCRIPTION:
Rationale why study should be conducted: Leiomyomas are the most common benign neoplasm in women; it has been estimated that these tumors occur in at least 25% of all women, which is probably an underestimation, because this figure is based on a select population. They are histologically composed by smooth muscle cells with bland, uniform, cigar-shaped nuclei that are arranged in interlacing bundles, showing little or no mitotic activity. Cellular leiomyomas (CLs) are described as leiomyomas that are significantly more cellular than the surrounding myometrium, often with crowding and overlapping of nuclei.

The presenting symptoms do not differ from those of patients with typical leiomyomas. On gross examination, CLs are more often soft and appear more tan or yellow and less circumscribed than the usual leiomyomas.

Pre-operatively, anyway, CLs can be recognized at ultrasound evaluation because they appear as hypoechoic uterine lesions. It has been demonstrated that patients with hypoechoic myoma have a significantly longer surgery time after treatment with a GnRH analog than for the rest of the pretreated fibroids or the untreated patients with hypoechoic myomas. Considering the predominant relevance of the traction maneuvers in laparoscopic myomectomy, the difficulty in adequately grasping the tumor is the key element in the longer operative time. The greater softening of the fibroid tissue is probably related to degenerative changes induced by the GnRH-analog pretreatment, particularly in those fibroids without an adequate fibrous "skeleton" and thus with the appearance as hypoechoic at the admission ultrasonography. From a pathologic point of view, these fibroids, when pretreated, showed a predominance of areas of coagulative necrosis and mixoid degeneration, causing longer operative time and showing unequivocally the negative effect of preoperative GnRH analog treatment for these kinds of uterine fibroids.

At the same time, hypoechoic CLs should be more responsive to ulipristal acetate treatment than common leiomyomas, given its antiproliferative activity in cultured leiomyoma cells.

The antiproliferative ulipristal effect, moreover, induces a condition of apoptotic necrosis that, compared to GnRH-a myxoid necrosis, probably allows an easier surgical enucleation of the tumor.

ELIGIBILITY:
Inclusion Criteria:

* hypoechoic uterine leiomyoma (echogenicity <3),
* intramural leiomyomas with an ultrasonographic size <20 cm but >4cm,
* indication to surgery (symptoms of menometrorrhagia,
* menstrual disorder,
* infertility,
* pelvic pain or pelvic pressure

Exclusion Criteria:

* submucosal leiomyoma,
* endometrial hyperplasia with atypia,
* history of uterine surgery

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Operative time (minutes) | At the time of skin closure at the end of the myomectomy
  To evaluate the difference in terms of operative times in patients with hypoechoic CLs submitted to laparoscopic myomectomy and preoperatively treated by ulipristal acetate or GnRh-a .

SECONDARY OUTCOMES:
Difficulty of leiomyoma enucleation assessed by surgeon on a VAS scale | Within 2 hours after the end of the myomectomy
  To compare surgical feasibility (VAS) in patients treated with Ulipristal Acetate and GnRH-a.
Intraoperative blood loss (delta Hb) | The day before surgery and 3 hours after the myomectomy
  To compare blood loss (delta HB) in patients treated with Ulipristal Acetate and GnRH-a.
Post-operative evaluation of leiomyomas characteristics | At the time of pathological assessment
  This is a composite outcome aimed to compare pathological myoma characteristics (cellularity, necrosis, fibrosis) in patients treated with Ulipristal Acetate and GnRH-a.

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Zullo, MD,PhD, Study Director — Magna Graecia University of Catanzaro; Roberta Venturella, Principal Investigator — Magna Graecia University of Catanzaro
Locations (1):
- Azienda Ospedaliera Pugliese-Ciaccio, Catanzaro, Catanzaro, Italy